CLINICAL TRIAL: NCT00660257
Title: Safety and Immunogenicity of Booster Dose of An Inactivated,Adjuvanted Whole-Virion Pandemic Influenza (H5N1)Vaccine in Two-Dose Primed Healthy Adults: A Single Center, Non-Randomized Clinical Trial
Brief Title: Safety and Immunogenicity of Booster Dose of An Inactivated,Adjuvanted Whole-Virion Pandemic Influenza(H5N1)Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Collaborators: Centers for Disease Control and Prevention, China (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-PanFlu-1002
Record Dates: First submitted 2008-04-15; First posted 2008-04-17 (Estimated); Last update posted 2008-04-17 (Estimated); Status verified 2008-04

CONDITIONS: Pandemic Influenza Vaccine; Prevention; Pandemic Influenza

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- No.1: 1.25 ug (Experimental)
  Interventions: Biological: pandemic influenza vaccine (H5N1 strain NIBRG-14)
- No.2: 2.5 ug (Experimental)
  Interventions: Biological: pandemic influenza vaccine (H5N1 strain NIBRG-14)
- No.3: 5.0 ug (Experimental)
  Interventions: Biological: pandemic influenza vaccine (H5N1 strain NIBRG-14)
- No. 4: 10 ug (Experimental)
  Interventions: Biological: pandemic influenza vaccine (H5N1 strain NIBRG-14)

INTERVENTIONS:
Biological: pandemic influenza vaccine (H5N1 strain NIBRG-14) — pandemic influenza vaccine (H5N1 strain NIBRG-14) booster (third) dose: 1.25 ug per dose, intramuscular injection
  Arms: No.1: 1.25 ug
Biological: pandemic influenza vaccine (H5N1 strain NIBRG-14) — pandemic influenza vaccine (H5N1 strain NIBRG-14) booster (third) dose: 2.5 ug per dose, intramuscular injection
  Arms: No.2: 2.5 ug
Biological: pandemic influenza vaccine (H5N1 strain NIBRG-14) — pandemic influenza vaccine (H5N1 strain NIBRG-14) booster (third) dose: 5.0 ug per dose, intramuscular injection
  Arms: No.3: 5.0 ug
Biological: pandemic influenza vaccine (H5N1 strain NIBRG-14) — pandemic influenza vaccine (H5N1 strain NIBRG-14) booster (third) dose: 1.25 ug per dose, intramuscular injection
  Arms: No. 4: 10 ug

SUMMARY:
A single center, non-randomized clinical trial in two-dose primed healthy adults to evaluate the safety and immunogenicity of a booster dose of an inactivated pandemic influenza (H5N1) vaccine (whole-virion, aluminium-adjuvanted).

ELIGIBILITY:
Inclusion Criteria:

* Had received two-dose priming vaccination in previous phase I trial
* Be able to show legal identity card for the sake of recruitment
* Be able to understand and sign the informed consent.

Exclusion Criteria:

* Woman： Who breast-feeding or planning to become pregnant during the study
* Any history of allergic reactions to vaccines or eggs
* Autoimmune disease or immunodeficiency
* Diabetes mellitus (type I or II), with the exception of gestational diabetes
* Serious angioedema episodes within the previous 3 years or requiring medication in the previous two years
* Hypertension that was not well controlled by medication or is more than 145/95 mmHg at enrollment
* Active malignancy or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of study
* Guillain-Barre Syndrome
* Women subjects with positive urinary pregnancy test
* Any history of immunosuppressive medications or cytotoxic medications or inhaled corticosteroids within the past six months
* History of any blood products administration within 3 months before the dosing
* Administration of any other investigational research agents within 30 days before the dosing
* Administration of any live attenuated vaccine within 30 days before the dosing
* Administration of subunit or inactivated vaccines, e.g. pneumococcal vaccine, or allergy treatment with antigen injections, within 14 days before the dosing
* Be receiving anti-TB prophylaxis or therapy currently
* Axillary temperature >37.0 centigrade at the time of dosing
* Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder requiring therapy that has not been well controlled on medication for the past two years; disorder requiring lithium; or suicidal ideation occurring within five years prior to enrollment
* Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent.

Ages: 19 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2007-01; Primary Completion 2007-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
HI antibody Neutralization antibody | 15 and 30 days after the booster dose

SECONDARY OUTCOMES:
local adverse reactions systemic adverse reactions temperature | 3 days after booster dose

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Lin JT, Li CG, Wang X, Su N, Liu Y, Qiu YZ, Yang M, Chen JT, Fang HH, Dong XP, Yin WD, Feng ZJ. Antibody persistence after 2-dose priming and booster response to a third dose of an inactivated, adjuvanted, whole-virion H5N1 vaccine. J Infect Dis. 2009 Jan 15;199(2):184-7. doi: 10.1086/595832. PMID 19067606